CLINICAL TRIAL: NCT03439384
Title: TEC4Home: Telehealth for Emergency-Community Continuity of Care Connectivity Via Home-Telemonitoring
Brief Title: TEC4Home Heart Failure: Using Home Health Monitoring to Support the Transition of Care
Acronym: TEC4Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kendall Ho, Lead, Digital Emergency Medicine; Professor, Department of Emergency Medicine, Faculty of Medicine, UBC, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-02846
Record Dates: First submitted 2018-01-16; First posted 2018-02-20 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A stepped wedge trial design was used to cluster and randomize recruiting sites into a schedule as to when sites would enroll participants into the control or intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Home Telemonitoring (Experimental): Patients will receive home telemonitoring equipment and monitor their health for 60 days post-enrollment. A monitoring nurse will receive and review the patients health data on a daily basis for the 60 day duration and provide remote care, counseling and education.
  Interventions: Device: Home Telemonitoring
- Control: No Home Telemonitoring (No Intervention): The patient will not receive any home telemonitoring once enrolled and will continue to receive the usual care he/she can expect as part of his/her care plan.

INTERVENTIONS:
Device: Home Telemonitoring — Patients will monitor their weight, blood pressure, oxygen saturation and symptoms with sensors and a tablet computer provided to them. Patients are asked to do this everyday for 60-days. A monitoring nurse will be receiving the data electronically and reviewing on a daily basis.
  Arms: Experimental: Home Telemonitoring

SUMMARY:
TEC4Home Heart Failure is a randomized controlled trial (RCT) that examines how home health monitoring (HHM) can support Heart Failure (HF) patients during the transition of care from hospital to home. The HHM solution includes a weight scale, blood pressure cuff, pulse oximeter and tablet computer, which patients use daily for 60 days to record these metrics and answer questions on their symptoms. This data is sent to a nurse who is able to monitor the patient's condition remotely. The hypothesis is that the TEC4Home HHM solution will be a cost-effective strategy to decrease 90-day Emergency Department (ED) revisits and hospital admission rates, and improve quality of life and self-management for patients living with Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Be 19 years of age or older (age of majority in British Columbia)
* Have one or more typical symptoms of Heart Failure (i.e. dyspnoea at rest or minimal exertion (includes orthopnoea, reduced exercise tolerance)) AND
* Have one or more typical signs of Heart Failure (i.e. elevated jugular venous pressure, pulmonary crepitations, pleural effusions, peripheral oedema) AND
* Have one or more objective measures of heart failure:
* Radiological congestion.
* Elevated BNP ≥ 400 pg/mL or NT-proBNP ≥ 1000 pg/mL.
* Reduced left ventricular ejection fraction <40% (or <45%) in previous 12 months.
* Diastolic dysfunction including tissue Doppler E/e' ratio > 15 in previous 12 months.
* Pulmonary capillary wedge pressure >20 mmHg.
* Diuretic therapy. The additional value of diuretic therapy (IV or oral) is debatable, as presumably unlikely (or unsafe) that patient with genuine HF will be discharged without diuretic.

Exclusion Criteria:

* Physical barriers e.g. unable to stand on scales.
* Cognitive impairment (e.g. MMSE <20), unless suitable caregiver support.
* Language (must be able to read and understand English), unless suitable caregiver support.
* Documented history of current and active substance misuse (within 3 months).
* Lack digital connectivity or landline phone connection.
* No regular care provider e.g. GP, or at least regular walk-in clinic.
* Existing intensive system of care: LVAD, transplant, dialysis.
* Anticipated improvement due to revascularization (PCI/CABG) or valve intervention during index hospitalization.
* Anticipated survival <90 days. Active palliative care, less-than level III care, disseminated malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of emergency department visits 90 days pre to 90 days post enrollment. | 90 days
  Hospital administrative data will be reviewed to assess the change in the number of emergency department visits 90 day pre to 90 days post enrollment and between study groups.
Change in the number of hospitalizations 90 days pre to 90 days post enrollment. | 90 days
  Hospital administrative data will be reviewed to assess the number of hospitalizations 90 day pre and 90 days post enrollment and between study groups.
Change in the length (in days) of hospital stays 90 days pre to 90 days post enrollment. | 90 days
  Hospital administrative data will be reviewed to assess the change in length of stay (measured in days) 90 day pre and 90 days post enrollment and between study groups.
Mortality rate | 90 days
  Administrative will be reviewed to determine the number of participants who passed away between study groups.

SECONDARY OUTCOMES:
Difference in quality of life (general) scores as assessed by the EuroQol- 5 Dimension Survey (EQ-5D). | 90 days
  A 5 item generic health-related quality of life questionnaire to be administered to all participants for comparison pre-post enrollment and between study groups.
Difference in quality of life (HF-specific) scores as assessed by the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ-12) scale. | 90 days
  A 12 item disease-specific quality of life questionnaire will be administered to all participants for comparison pre-post enrollment and between study groups.
Difference in self-care efficacy scale scores as assessed by the European Heart Failure Self-care Behaviour Scale. | 90 days
  A 9 item scale to asses a patient's self-care behaviours and attitudes specific to Heart Failure will be administered to all participants for comparison pre-post enrollment and between study groups.
Difference in costs and savings via administrative data and a self-report healthcare utilization survey. | 90 days
  Costs related to healthcare utilization and other health-related out of pocket and system costs will be assessed and compared 90 days pre to 90 days post enrollment and between study groups.
Impact on communication between healthcare providers and patients via surveys. | 90 days
  Surveys about end-user experience will be used to collect feedback from patient participants, nurses and other healthcare providers involved to understand the impact of home health monitoring on communication during the transition of care.
Impact on communication between healthcare providers and patients via interviews. | 90 days
  Interviews about end-user experience will be used to collect feedback from patient participants, nurses and other healthcare providers involved to understand the impact of home health monitoring on communication during the transition of care.

CONTACTS AND LOCATIONS:
Overall Officials: Kendall Ho, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- UBC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ho K, Novak Lauscher H, Cordeiro J, Hawkins N, Scheuermeyer F, Mitton C, Wong H, McGavin C, Ross D, Apantaku G, Karim ME, Bhullar A, Abu-Laban R, Nixon S, Smith T. Testing the Feasibility of Sensor-Based Home Health Monitoring (TEC4Home) to Support the Convalescence of Patients With Heart Failure: Pre-Post Study. JMIR Form Res. 2021 Jun 3;5(6):e24509. doi: 10.2196/24509. PMID 34081015